CLINICAL TRIAL: NCT06558786
Title: Prospective Registry Study of Multimodality Therapy for Oligometastatic Adenocarcinoma of the Esophagus or Gastroesophageal Junction
Brief Title: Registry for Esophageal and Gastroesophageal Junction Cancer
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 24-206
Record Dates: First submitted 2024-08-13; First posted 2024-08-19 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Gastroesophageal-junction Cancer; Esophageal Cancer
Keywords: Quality-of-Life Assessments; 24-206
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Esophageal and Gastroesophageal Junction Cancer: Patients will undergo assessment with the EORTC QLQ-C30 and QLQ-OGS25 questionnaires. Those patients who undergo local therapy will occur at baseline, months 7-9 within 45 days of local therapy, and one year/time of progression. Those patients who do not undergo local therapy will undergo assessment at baseline, at 6 months, and at one year.
  Interventions: Other: EORTC QLQ-C30 questionnaire; Other: QLQ-OGS25 questionnaire

INTERVENTIONS:
Other: EORTC QLQ-C30 questionnaire — The EORTC QLQ-C30 has 30 items arranged into 9 scales and 6 single items. The scales are divided into 5 function scales (physical, role, cognitive, emotional, and social function), 3 symptom scales (fatigue, pain, and nausea or vomiting), and 1 global health status/quality-of-life scale. The 6 single items address specific symptoms (dyspnea, appetite loss, insomnia, constipation, and diarrhea) and the financial impact of the disease. Each item has 4 response alternatives: (1) "not at all," (2) "a little," (3) "quite a bit," and (4) "very much," except for the global health status/quality-of-life scale, which has response options ranging from (1) "very poor" to (7) "excellent." For analysis, all questionnaire responses will be transformed into scores on a linear scale of 0 to 100 in accordance with the EORTC scoring manual. Mean scores with standard deviations will be calculated, with a higher score indicating a better health-related quality of life.
Other: QLQ-OGS25 questionnaire — The QLQ-OGS25 is specific for esophageal, GEJ, or gastric cancer and consists of a symptom scale only. The QLQ-OGS25 has 6 scales: dysphagia, eating restrictions, reflux, odynophagia, pain, and anxiety. Scales have good reliability (α range, 0.67-0.87), and they distinguish between tumor sites and disease stage. The response format is a 4-point Likert scale. Responses to the questionnaires will be transformed into a scale of 0 to 100 using the EORTC guidelines, with a higher score indicating a deterioration of symptoms.

SUMMARY:
The purpose of this registry study is to create a database-a collection of information-for better understanding standard treatments for esophageal and Gastroesophageal Junction Cancer/GEJ cancer. Researchers will use the information from this database to learn more about the effectiveness of different treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed stage IV adenocarcinoma of the esophagus or GEJ with OMD at the time of diagnosis, defined as the following:
* Retroperitoneal lymph nodes (e.g., para-aortal, intra-aorto-caval, parapancreatic, or mesenterial lymph node)
* Liver
* Lung
* Extra-abdominal lymph nodes (e.g., supraclavicular or cervical lymph nodes)
* Adrenal gland
* Unilateral or bilateral ovarian metastases (in the absence of gross or microscopic peritoneal disease [positive cytology])
* Bone
* ≤2 sites of disease (excluding the primary tumor and regional lymph nodes)
* ≤3 tumors within each organ system
* ≤5 metastases
* All nonregional lymph nodes (including cervical, supraclavicular, and retroperitoneal nodal disease) are considered 1 discrete lesion
* Satellite lesions in the primary esophageal malignancy, such as skipped esophageal primaries, are not considered metastatic sites
* All sites of disease must be amenable to complete local therapy after systemic therapy, according to the treating physician. Treatment modalities include:
* Surgery
* Definitive chemoradiation
* Stereotactic radiation
* Ablation or similar techniques (e.g., irreversible electroporation)
* Age ≥18 years

Exclusion Criteria:

* Presence of metastases, at the time of diagnosis, to the following:

  * Peritoneum, including positive peritoneal lavage (on the basis of baseline diagnostic laparoscopy to rule out gross disease and positive peritoneal lavage cytology; laparoscopy may be omitted for patients in whom all sites of disease are above the diaphragm)
  * Malignant pleural effusion
  * Brain metastases or leptomeningeal disease
  * Other sites not specifically noted must be reviewed and approved by the PIs
  * Any site of disease that is not amenable to definitive local therapy
* Unfit for best systemic therapy
* Metachronous OMD
* Secondary primary cancer, with the exclusion of basal cell carcinoma of the skin
* Pregnant, lactating, or intending to become pregnant
* Unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at MSK.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2029-08-12 (Estimated); Study Completion 2029-08-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 1 year
  Estimate 12-month PFS among patients who undergo definitive local therapy after induction chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Molena, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm